CLINICAL TRIAL: NCT04498663
Title: Emotion- and Relationship-Focused Therapeutic Interview for Chronic Musculoskeletal Pain: A Randomized Trial
Brief Title: The Pain & Stress Interview Study for People With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark A. Lumley (Other)
Responsible Party: Sponsor-Investigator, Mark A. Lumley, Distinguished Professor of Psychology, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20-04-2070
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Musculoskeletal Pain
Keywords: Chronic Pain
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at a 1:1 ratio to one of two groups--either the therapeutic interview condition or the waitlist control condition.
Masking Description: Both patient and research assistant interviewer will be blinded to condition assignment during the baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Interview Condition (Experimental): The therapeutic interview for chronic pain will be a one-session interview lasting approximately 90 minutes. The goals of the therapeutic interview are to promote awareness of the role of trauma and interpersonal stress in pain, to encourage experience of emotions associated with interpersonal stressors and conflicts, and to encourage more adaptive interpersonal communication in current relationships.
  Interventions: Behavioral: Emotion- and Relationship-Focused Therapeutic Interview
- Waitlist Control Condition (No Intervention): Participants in the waitlist control condition will receive a delayed interview (after 6-week follow-up assessment), if they choose to do so.

INTERVENTIONS:
Behavioral: Emotion- and Relationship-Focused Therapeutic Interview — In this study, the therapeutic interview will be one-session lasting 90 minutes. Participants will explore prior and ongoing stressful life experiences. Participants will be educated about the role of stress in pain and will be encouraged to identify links between stressors, psychological and emotional conflicts related to the stressors, and their pain symptoms. The interview will encourage the experience and expression of previously avoided emotions related to interpersonal stressors.
  Arms: Therapeutic Interview Condition

SUMMARY:
The goal of the study is to determine whether a brief, therapeutic interview can help patients improve their pain and health by addressing psychological issues that are known to drive chronic musculoskeletal pain. This randomized, controlled trial tests the efficacy of a brief, one-session therapeutic interview for patients with chronic musculoskeletal pain and histories of childhood adversity. Adults with chronic musculoskeletal pain will be randomized to either a therapeutic interview condition or a waitlist control condition. The therapeutic interview will be 90-minute session during which participants will be encouraged to disclose stressful experiences, express important emotions, and identify connections between their life stress and their pain, which we hope will increase their psychological attributions for pain and reduce their pain, interpersonal problems, and psychological distress. The study will compare the therapeutic interview condition to a delayed interview condition and will follow patients for 6 weeks to identify changes in response to the interview. Participants in the therapeutic interview condition are expected to show more improvement on pain severity, pain interference, psychological distress, interpersonal function, and psychological attitudes toward pain at follow-up, relative to participants in the delayed interview condition.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to test the efficacy of a brief, one-session therapeutic interview for patients who are seeking biomedical care for their chronic musculoskeletal pain and who also have self-reported trauma histories. Participants will be randomized to either a therapeutic interview condition or a waitlist control condition and and will follow patients for 6 weeks to identify health and attitude changes in response to the interview.

This study will recruit adults with chronic musculoskeletal pain and reported histories of childhood adversity. Participants will be adults with primary musculoskeletal pain such as low back pain, neck pain, and fibromyalgia. In addition, only those patients who also report a significant history of childhood adversity will be eligible for this study, as determined by a score of 3 or higher on the Adverse Childhood Experiences (ACE) Scale. Patients will be excluded if they: a) have a current psychotic disorder or b) are unable to communicate in English, or c) are scheduled for an upcoming surgery within the next 2 months. Participants will be allowed to engage in this study regardless of current medication use or engagement in other treatment.

Patients who are interested in participating will complete a brief online screening to determine eligibility and will be provided with basic information about the study. Once consented, baseline measures will be completed online, and participants will be randomized, 1:1, to the therapeutic interview condition or waitlist control condition. Those who are randomized to the therapeutic interview condition will complete their interview as soon as possible after completing baseline measures. The interview will be conducted either in-person at the Stress & Health Laboratory at Wayne State University, or remotely via a secure telehealth platform (depending on COVID-19 restrictions). Follow-up measures will be administered at 6 weeks after the interview (or at the equivalent time for the waitlist group). Participants in the waitlist control condition will be given the opportunity to receive the therapeutic interview after completion of the follow-up measures.

The therapeutic interview will be a one-session interview lasting approximately 90 minutes. The interview will be conducted by trained interviewers (i.e., clinical psychology graduate students). The goals of the therapeutic interview are to promote awareness of the role of trauma and interpersonal stress in pain, to encourage experience of emotions associated with interpersonal stressors and conflicts, and to encourage more adaptive interpersonal communication in current relationships. The interview has five primary components. The first component involves eliciting a brief pain history from the participants. The next component explores participants' stressful life experiences, including those that occurred during their childhood and those that might be affecting their current life. The next component will introduce participants to a model of emotions that illustrates how suppressing important, healthy feelings in relationships can lead to symptoms (e.g. anxiety, pain, stress). Participants will be encouraged to identify the feelings that are most difficult for them to express in relationships and the ways in which avoiding these feelings leads to prolonged stress or worse pain. The next component involves encouraging participants to identify key, conflictual relationships and to express their previously avoided, healthy feelings (e.g. assertion, tenderness, grief). The final and 5th component will explore how the interview affected their beliefs about the role of stress and emotions in pain. The interviewer will provide a summary of their strengths and areas for improvement related to their emotions and interpersonal functioning.

There will be clinical outcomes that reflect changes in pain severity and pain interference, pain-related anxiety, and emotional distress. There will be behavioral outcomes that capture changes in patients' interpersonal assertiveness, substance use, and adaptive affective functioning (defined as one's cognitive, behavioral, and emotional responses to one's healthy feelings or needs). Finally, there will be attitudinal outcomes that reflect changes in patients' attributions about the role of psychological and brain-based factors in pain.

ELIGIBILITY:
Inclusion Criteria:

* a chronic primary musculoskeletal pain condition
* significant history of childhood adversity (score of 3 or higher on the Adverse Childhood Experiences (ACE) Scale.

Exclusion Criteria:

* current psychotic disorder
* unable communicate in English
* unable to read
* surgery scheduled within 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pain severity from baseline to 6-week follow-up | 6-week follow-up
  Brief Pain Inventory pain severity scale (0 - 10; higher values = greater pain severity)

SECONDARY OUTCOMES:
Change in pain interference from baseline to 6-week follow-up | 6-week follow-up
  Brief Pain Inventory pain interference scale (0 - 10; higher values = greater pain interference)
Change in pain anxiety from baseline to 6-week follow-up | 6-week follow-up
  Pain Anxiety Symptom Scale-20 (sum ranges from 0 to 100; higher values = greater pain anxiety
Change in anxiety from baseline to 6-week follow-up | 6-week follow-up
  PROMIS anxiety scale (0 to 4; higher values = greater anxiety)
Change in depression from baseline to 6-week follow-up | 6-week follow-up
  PROMIS depression scale (0 to 4; higher values = greater depression)
Change in anger from baseline to 6-week follow-up | 6-week follow-up
  PROMIS anger scale (0 to 4; higher values = greater anger)
Change in pain attributions to psychological processes from baseline to 6-week follow-up | 6-week follow-up
  Pain attributions psychological subscale (0 to 4; higher values = greater psychological attribution)
Change in pain attributions to brain processes from baseline to 6-week follow-up | 6-week follow-up
  Pain attributions brain subscale (0 to 4; higher values = greater brain attributions)
Change in pain beliefs (harm, control, emotion) from baseline to 6-week follow-up | 6-week follow-up
  Survey of Pain Attitudes subscales (1 to 5; higher values = stronger beliefs)

OTHER OUTCOMES:
Change in alcohol use frequency from baseline to 6-week follow-up | 6-week follow-up
  Alcohol use item (1 to 7; higher = greater alcohol use)
Change in pain medication use from baseline to 6-week follow-up | 6-week follow-up
  Item assessing pain medication use (1 to 5; higher = greater medication use)
Change in affect phobia from baseline to 6-week follow-up | 6-week follow-up
  Affect Phobia Test (1 to 5; lower values = affect phobia)
Change in assertiveness from baseline to 6-week follow-up | 6-week follow-up
  Rathus Assertiveness Schedule short form (- 3 to + 3; higher values = greater assertion)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lumley, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University Department of Psychology, Detroit, Michigan, United States

REFERENCES:
- [Derived] Krohner S, Town J, Cannoy CN, Schubiner H, Rapport LJ, Grekin E, Lumley MA. Emotion-Focused Psychodynamic Interview for People with Chronic Musculoskeletal Pain and Childhood Adversity: A Randomized Controlled Trial. J Pain. 2024 Jan;25(1):39-52. doi: 10.1016/j.jpain.2023.07.017. Epub 2023 Jul 20. PMID 37479050